CLINICAL TRIAL: NCT04055740
Title: Intravascular ultraSound (IVUS) Imaging During transvEnous Lead Extraction (ISEE)
Brief Title: Intravascular Ultrasound (IVUS) Imaging During Transvenous Lead Extraction
Acronym: ISEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-1600
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-08

CONDITIONS: Device Malfunction; ICD; Pacemaker Lead Dysfunction
Keywords: CIED

STUDY DESIGN:
Intervention Model Description: Single cohort of patients undergoing transvenous lead extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IVUS imaging (Experimental): IVUS imaging will be used each patient undergoing transvenous lead extraction to visualize ILA
  Interventions: Device: IVUS Imaging

INTERVENTIONS:
Device: IVUS Imaging — IVUS or radial-ICE (intracardiac echocardiography) is a visualization tool used in many cardiac procedures including electrophysiology procedures (catheter ablation). Its utility in identifying ILA will be assessed in this study.

SUMMARY:
The purpose of this study is to prospectively evaluate intravascular ultrasound (IVUS) imaging as a tool for grading the presence and characterization of intravascular lead adherence (ILA, or scarring) to cardiovascular implantable electronic device (CIED) leads during transvenous lead extraction (TLE) procedures in a multi-center study. IVUS should identify the location and severity of these adhesions, which the investigators will then correlate to difficulty of the extraction procedure using metrics like pulses of laser energy delivered and time required to traverse an area of fibrosis or ILA. The investigators will be focusing primarily on the section from innominate vein (INNV) down through the superior vena cava (SVC) to the right atrium.

Using IVUS to view blood vessels and the heart structure is approved by the Food and Drug Administration (FDA). Using it as described in this study is off label because of the manner in which it is advanced to the SVC, through the right atrium. While it is not restricted from use in this way, it is not specifically on-label. It should be noted that the use of IVUS during TLE procedures as proposed in this study is routine at the University of Chicago and patients will undergo this procedure regardless of participation in this study. The EP physician team regards the use of IVUS during TLE to be nonsignificant risk.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 21 years of age
* Patients with at least one lead over 1 year dwell time requiring extraction

Exclusion Criteria:

* Inability of patient capacity to provide consent for themselves either due to medical or psychiatric comorbidity
* Venous occlusion to the extent that the IVUS catheter cannot pass
* Leads < 1 year dwell time requiring extraction

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hemal Nayak, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greenspon AJ, Patel JD, Lau E, Ochoa JA, Frisch DR, Ho RT, Pavri BB, Kurtz SM. 16-year trends in the infection burden for pacemakers and implantable cardioverter-defibrillators in the United States 1993 to 2008. J Am Coll Cardiol. 2011 Aug 30;58(10):1001-6. doi: 10.1016/j.jacc.2011.04.033. PMID 21867833
- [Background] Mond HG, Irwin M, Ector H, Proclemer A. The world survey of cardiac pacing and cardioverter-defibrillators: calendar year 2005 an International Cardiac Pacing and Electrophysiology Society (ICPES) project. Pacing Clin Electrophysiol. 2008 Sep;31(9):1202-12. doi: 10.1111/j.1540-8159.2008.01164.x. PMID 18834475
- [Background] Joy PS, Kumar G, Poole JE, London B, Olshansky B. Cardiac implantable electronic device infections: Who is at greatest risk? Heart Rhythm. 2017 Jun;14(6):839-845. doi: 10.1016/j.hrthm.2017.03.019. Epub 2017 Mar 16. PMID 28315744
- [Background] Kusumoto FM, Schoenfeld MH, Wilkoff BL, Berul CI, Birgersdotter-Green UM, Carrillo R, Cha YM, Clancy J, Deharo JC, Ellenbogen KA, Exner D, Hussein AA, Kennergren C, Krahn A, Lee R, Love CJ, Madden RA, Mazzetti HA, Moore JC, Parsonnet J, Patton KK, Rozner MA, Selzman KA, Shoda M, Srivathsan K, Strathmore NF, Swerdlow CD, Tompkins C, Wazni O. 2017 HRS expert consensus statement on cardiovascular implantable electronic device lead management and extraction. Heart Rhythm. 2017 Dec;14(12):e503-e551. doi: 10.1016/j.hrthm.2017.09.001. Epub 2017 Sep 15. No abstract available. PMID 28919379
- [Background] Brunner MP, Cronin EM, Wazni O, Baranowski B, Saliba WI, Sabik JF, Lindsay BD, Wilkoff BL, Tarakji KG. Outcomes of patients requiring emergent surgical or endovascular intervention for catastrophic complications during transvenous lead extraction. Heart Rhythm. 2014 Mar;11(3):419-25. doi: 10.1016/j.hrthm.2013.12.004. Epub 2013 Dec 4. PMID 24315967
- [Background] Bracke F. Complications and lead extraction in cardiac pacing and defibrillation. Neth Heart J. 2008 Oct;16(Suppl 1):S28-31. PMID 18958266
- [Background] Mazzone P, Tsiachris D, Marzi A, Ciconte G, Paglino G, Sora N, Sala S, Vergara P, Gulletta S, Della Bella P. Predictors of advanced lead extraction based on a systematic stepwise approach: results from a high volume center. Pacing Clin Electrophysiol. 2013 Jul;36(7):837-44. doi: 10.1111/pace.12119. Epub 2013 Mar 19. PMID 23510021
- [Background] Maytin M, Epstein LM, John RM. Lead implant duration does not always predict ease of extraction: extraction sheath may be required at < 1 year. Pacing Clin Electrophysiol. 2011 Dec;34(12):1615-20. doi: 10.1111/j.1540-8159.2011.03225.x. Epub 2011 Oct 20. PMID 22017453
- [Background] Enriquez A, Saenz LC, Rosso R, Silvestry FE, Callans D, Marchlinski FE, Garcia F. Use of Intracardiac Echocardiography in Interventional Cardiology: Working With the Anatomy Rather Than Fighting It. Circulation. 2018 May 22;137(21):2278-2294. doi: 10.1161/CIRCULATIONAHA.117.031343. PMID 29784681
- [Background] Bongiorni MG, Di Cori A, Soldati E, Zucchelli G, Arena G, Segreti L, De Lucia R, Marzilli M. Intracardiac echocardiography in patients with pacing and defibrillating leads: a feasibility study. Echocardiography. 2008 Jul;25(6):632-8. doi: 10.1111/j.1540-8175.2008.00656.x. PMID 18652009
- [Background] Sadek MM, Cooper JM, Frankel DS, Santangeli P, Epstein AE, Marchlinski FE, Schaller RD. Utility of intracardiac echocardiography during transvenous lead extraction. Heart Rhythm. 2017 Dec;14(12):1779-1785. doi: 10.1016/j.hrthm.2017.08.023. Epub 2017 Aug 24. PMID 28843419
- [Background] Santoshi RKN, Lakhanpal S, Satwah V, Lakhanpal G, Malone M, Pappas PJ. Iliac vein stenosis is an underdiagnosed cause of pelvic venous insufficiency. J Vasc Surg Venous Lymphat Disord. 2018 Mar;6(2):202-211. doi: 10.1016/j.jvsv.2017.09.007. Epub 2017 Dec 29. PMID 29292119
- [Background] Ganguli S, Hawkins BM, Abtahian F, Abu-Fadel MS, Walker TG, MacKay C, Jaff MR, Weinberg I. Comparison of Inferior Vena Cava Filters Placed at the Bedside via Intravenous Ultrasound Guidance Versus Fluoroscopic Guidance. Ann Vasc Surg. 2017 Feb;39:250-255. doi: 10.1016/j.avsg.2016.06.013. Epub 2016 Aug 28. PMID 27581130
- [Background] Kassavin DS, Constantinopoulos G. The transition to IVUS-guided IVC filter deployment in the nontrauma patient. Vasc Endovascular Surg. 2011 Feb;45(2):142-5. doi: 10.1177/1538574410393753. Epub 2011 Jan 28. PMID 21278179
- [Background] Jeyabalan G, Wallace JR, Chaer RA, Leers SA, Marone LK, Makaroun MS. Endovascular strategies for treatment of embolizing thoracoabdominal aortic lesions. J Vasc Surg. 2014 May;59(5):1256-64. doi: 10.1016/j.jvs.2013.11.068. Epub 2014 Jan 14. PMID 24433783
- [Background] Di Valentino M, Alerci M, Bogen M, Tutta P, Sartori F, Marty B, von Segesser L, Gallino A. Telementoring during endovascular treatment of abdominal aortic aneurysms: a prospective study. J Endovasc Ther. 2005 Apr;12(2):200-5. doi: 10.1583/04-1421.1. PMID 15823067
- [Background] Kolluri R, Fowler B, Ansel G, Silver M. A novel duplex finding of superficial epigastric vein flow reversal to diagnose iliocaval occlusion. J Vasc Surg Venous Lymphat Disord. 2017 May;5(3):358-362. doi: 10.1016/j.jvsv.2017.01.017. PMID 28411703
- [Background] Lewis RK, Pokorney SD, Greenfield RA, Hranitzky PM, Hegland DD, Schroder JN, Lin SS, Milano C, Daubert JP, Smith PK, Hurwitz LM, Piccini JP. Preprocedural ECG-gated computed tomography for prevention of complications during lead extraction. Pacing Clin Electrophysiol. 2014 Oct;37(10):1297-305. doi: 10.1111/pace.12485. Epub 2014 Sep 8. PMID 25195955
- [Background] Biefer HR, Hurlimann D, Grunenfelder J, Salzberg SP, Steffel J, Falk V, Starck CT. Generator pocket adhesions of cardiac leads: classification and correlation with transvenous lead extraction results. Pacing Clin Electrophysiol. 2013 Sep;36(9):1111-6. doi: 10.1111/pace.12184. Epub 2013 May 28. PMID 23713912

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment closed across the study due to low enrollment.
Period: Overall Study
Arm/Group | IVUS Imaging
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IVUS Imaging
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants] — One patient had missing age. Population: One patient had missing age.
  Participants
    number analyzed (Participants) | 30
    <=18 years | 0
    Between 18 and 65 years | 18
    >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient had missing age.
  years
    number analyzed (Participants) | 30
    (all) | 63.6 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient had missing sex.
  Participants
    number analyzed (Participants) | 30
    Female | 15
    Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 2 patients did not have data to determine BMI.
  kg/m^2
    number analyzed (Participants) | 29
    (all) | 29.68 (6.29)
Height [Mean (Standard Deviation); unit: cm] — Population: One patient had missing height.
  cm
    number analyzed (Participants) | 30
    (all) | 170.2 (12.64)

OUTCOME MEASURES:

1. Primary Outcome: IVUS Grades
Description: Operators will be able to successfully grade the degree of intravascular lead adherence (ILA) seen using IVUS imaging.
  Using the following scale, grading of ILA in each zone of interest, based on relative motion of lead will be performed:
  i. Grade 1: Freely mobile, Rarely adjacent to vasculature ii. Grade 2: Restricted mobility, Frequently adjacent to vasculature iii. Grade 3: Immobile, Always adjacent to vasculature iv. Grade L, added to number: Lead-to-lead binding
Time Frame: 6 hours
Population: 3 patients did not have any ILA grades.
Measure: Mean (Standard Deviation); unit: Grade
Arm/Group | IVUS Imaging
Number analyzed (Participants) | 28
Grade
  Right sided devices Zone1/2: number analyzed (Participants) | 3
  Right sided devices Zone1/2 | 1.33 (0.58)
  Right sided devices Zone 3: number analyzed (Participants) | 3
  Right sided devices Zone 3 | 1 (0)
  Left sided devices Zone 1: number analyzed (Participants) | 21
  Left sided devices Zone 1 | 1.57 (0.81)
  Left sided devices Zone 2: number analyzed (Participants) | 25
  Left sided devices Zone 2 | 1.44 (0.58)
  Left sided devices Zone 3: number analyzed (Participants) | 25
  Left sided devices Zone 3 | 1.32 (0.63)
  All devices, all zones | 1.40 (0.50)
Statistical Analysis 1: Comparison: IVUS Imaging; H0: rho = 0 Spearman correlation coefficient calculated between average ILA grade and total time of lead extraction; Test type: Superiority; p = 0.2201, Spearman Correlation Coefficient; This test measures correlation of avg ILA grade per patient with total time of lead extraction. Average ILA grade of all patients in outcome measures
Statistical Analysis 2: Comparison: IVUS Imaging; H0: rho = 0 Spearman Correlation coefficient calculated between average ILA grades and laser pulsations; Test type: Superiority; p = 0.5157, Spearman Correlation Coefficient; This measures correlation of avg ILA grade per patient with total laser pulsations used for extraction. Avg ILA grade of patients in outcome measures

2. Secondary Outcome: Extraction Difficulty Metrics
Description: Operators will record the energy and time necessary to traverse binding sites and will be able to correlate these two metrics to IVUS ILA grade
  Extraction difficulty was measured by correlating IVUS ILA grade to lead dwell time - the amount of time it took to extract the lead.
  Using the following scale, grading of ILA in each zone of interest, based on relative motion of lead was performed:
  i. Grade 1: Freely mobile, Rarely adjacent to vasculature ii. Grade 2: Restricted mobility, Frequently adjacent to vasculature iii. Grade 3: Immobile, Always adjacent to vasculature iv. Grade L, added to number: Lead-to-lead binding
Time Frame: Through study completion, expected to be 6 months
Population: Means calculated for patients with left sided devices vs patients with right sided devices - 4 patients had missing data
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IVUS Imaging
Number analyzed (Participants) | 28
minutes
  Right sided devices: number analyzed (Participants) | 2
  Right sided devices | 26.5 (21.92)
  Left sided devices: number analyzed (Participants) | 22
  Left sided devices | 34.91 (36.94)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | IVUS Imaging
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04055740/Prot_SAP_000.pdf